CLINICAL TRIAL: NCT06966622
Title: Comparison of Ngenuity and Traditional Microscopy in Assessing Retinal Function Recovery Post-ICL Surgery
Brief Title: Comparison of Retinal Damage in ICL Implantation Using 3D Visualization System vs. Microscope
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fuzhou Eye Hospital (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FZYKYY-KY-2025-002
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-05

CONDITIONS: High Myopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D visualization system (Experimental)
  Interventions: Procedure: 3D visualization system with coaxial illumination
- Microscope (Active Comparator)
  Interventions: Procedure: microscope with standard illumination

INTERVENTIONS:
Procedure: 3D visualization system with coaxial illumination — operation through 3D visualization system with coaxial illumination
  Arms: 3D visualization system
Procedure: microscope with standard illumination — operation through microscope with standard illumination
  Arms: Microscope

SUMMARY:
Implantable collamer lens (ICL) implantation is considered one of the most effective surgical treatments for high myopia. The procedure primarily involves adjusting the position of the ICL within the eye. However, precise calculation of the ICL optical power may cause the surgical light source to remain focused on the macular area during this process, potentially leading to iatrogenic light-induced damage. Theoretically, the combination of a 3D visualization surgical system and coaxial illumination technology can reduce the illumination intensity and decrease iatrogenic light damage. This study aims to compare the retinal physiological changes in patients undergoing ICL surgery through 3D visualization surgical system with coaxial illumination versus a traditional microscope with standard illumination.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of high myopic
* Aged 18-40 years
* Desire to improve their refractive status via ICL surgery
* Relatively stable refractive error (change ≤ 0.50 D per year for two consecutive years)
* Central anterior chamber depth ≥ 2.8 mm
* Open angles
* Corneal endothelial cell density ≥ 2000 cells/mm2.

Exclusion Criteria:

* Cataracts
* Corneal diseases,
* Glaucoma,
* Nystagmus,
* Strabismus,
* Lens subluxation,
* Severe vitreoretinal diseases,
* Other ocular diseases
* A history of ocular trauma
* A history of ocular surgery

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
b-wave amplitude | 1 day pre-op; 1 day post-op; 7 days post-op; 30 days post-op

SECONDARY OUTCOMES:
a-wave amplitude | 1 day pre-op; 1 day post-op; 7 days post-op; 30 days post-op
macular vessel density | 1 day pre-op; 1 day post-op; 7 days post-op; 30 days post-op
Uncorrected visual acuity | 1 day pre-op; 1 day post-op; 7 days post-op; 30 days post-op
Best-corrected visual acuity | 1 day pre-op; 1 day post-op; 7 days post-op; 30 days post-op

OTHER OUTCOMES:
Intraoperative illumination intensity | surgery beginning
Surgical time | Starting with the making of the surgical incision and ending with incision closure